CLINICAL TRIAL: NCT04005521
Title: Preventive Randomized Study Regarding Jaw- and Swallowing Intervention for Patients Receiving Radiotherapy for Head and Neck Cancer: the Effect of Preventive Intervention for Trismus, Swallowing Function and Quality of Life
Brief Title: Randomized Study Regarding Preventive Jaw- and Swallowing Intervention for Patients with Head and Neck Cancer
Acronym: HNC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lisa Tuomi, Principal Investigator, Vastra Gotaland Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00
Record Dates: First submitted 2019-06-13; First posted 2019-07-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Neoplasm; Trismus; Deglutition Disorders
MeSH Terms: conditions — Head and Neck Neoplasms; Trismus; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preventive intervention (Experimental): Patient will perform daily exercise: jaw and swallwing exercises, as well as are encouraged to eat and drink for as long as possible during treatment
  Interventions: Behavioral: Preventive intervention
- Control group (No Intervention): No intervention, only encouragement to eat and drink for as long as possible during treatment

INTERVENTIONS:
Behavioral: Preventive intervention — Preventive, structured exercise protocol
  Arms: Preventive intervention

SUMMARY:
The study includes patients with tumors of the oropharynx, larynx and hypopharynx scheduled to receive radiotherapy with curative intent (+/- chemotherapy). The patients will be randomized into either an intervention group (performing a preventive jaw- and swallowing exercise protocol before and during radiotherapy) or a control group no performing a exercise protocol. All patients will be encouraged to eat or drink for as long as possible during the therapy. All patients will meet with a speech-language therapist weekly during radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer (tumors of the oropharynx, pharynx, hypopharynx and larynx)
* Receiving radiohterpay (+/- chemotherapy) with curative intent
* No previous trismus or dysphagia

Exclusion Criteria:

* Surgery due to head and neck cancer
* Previous treatment for head and neck cancer
* Tracheostomized patients
* No teeth
* Inability to perform exercise intervention
* Inability to independently fill out questionnaires in Swedish
* Previous neurologic or neuromuscular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximal Interincisal opening (MIO) | 1 month post radiotherapy
  Jaw opening measured in millimeters. A MIO <36 mm is considered as trismus. i.e. limited jaw-opening.
Swallowing ability | 1 month after radiotherapy
  Swallowing ability measured with Functional Endoscopic Examination of Swallowing (FEES)

SECONDARY OUTCOMES:
Trismus and jaw related symptoms | Up to 5 years post radiotherapy
  Patient Reported Outcomes (PRO) measured with Gothenburg Trismus Questionnaire (GTQ). The GTQ consists of 21 items divided into 3 domains; Jaw related problems, Eating limitations and Muscular tension and eight single items concerning facial pain, limitations in mouth opening and inabilities to function on social and working contexts. The GTQ domains range from 0-100 where 0 equals to absence of symtoms and 100 equals worst possible symptoms.
Dysphagia related symtoms | Up to 5 years post radiotherapy
  PRO measured with M.D Anderson Dysphagia Inventory (MDADI). This is a cancer-specific instrument measuring dysphagia, social function and quality of life in head and neck cancer patients. It consists of 19 items in four domains; emotional, physical, functional and global quality of life. The range for each subscale is 20-100 where 100 indicates best possible swallowing, i.e. better outcome.
Health related quality of life (HRQL) | Up to 5 years post radiotherapy
  Measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) core questionnaire (c30). Consists of 30 items divided into six functional domains (Physical, Role, Cognitive, Emotional, and Social Functioning and Global Quality of life), three symptom scales (Fatigue, Pain, and Nausea/Vomiting) and six single items (Constipation, Diarrhea, Insomnia, Dyspnea, Appetite Loss, and Financial Difficulties). All domains range from 0-100. For the functional domains a higher score indicates good function, while for all other domains a high score indicates a high prevalence of symtoms, i.e. worse HRQL.
Health related quality of life (HRQL) | Up to 5 years post radiotherapy
  Measured with the EORTC QLQ Head and neck module (HN35). It consists of 35 questions regarding symptoms more specific to the head and neck cancer population, and domain scores range from 0-100, where a higher score represents the prevalence of more symtoms, i.e. worse HRQL.
Swallowing ability | Up to 5 years post radiotherapy
  Swallowing ability measured with FEES
Maximal Interincisal opening (MIO) | Up to 5 years post radiotherapy
  Jaw opening measured in millimeters

OTHER OUTCOMES:
Cost | Up to 5 years post radiotherapy
  The cost of intervention compared to usual care. Costs in Swedish crowns (SEK) for the intervention and all visits to healthcare during 5 years will be recorded.
Quality of life for cost-effectiveness analysis | Up to 5 years post radiotherapy
  The outcomes of intervention compared to usual care using European Quality of life 5 dimensions (EQ5D).
Quality Adjusted Life Years (QALY) | Up to 5 years post radiotherapy
  QALY is a measurement that combines health-related quality of life (HRQL) and life expectancy in one index. The index range between 0 and 1, where 0 equals death and 1 represents perfect health. Thus, 1 QALY corresponds to 1 year of perfect health. This is calculated using the EQ-5D.
Incremental Cost Effectiveness Ratio (ICER) | Up to 5 years post radiotherapy
  Incremental cost for each QALY for the intervention group will be calculated using a Markov model which combines the costs and EQ-5D. The ICER will then be compared to the maximum willingness to pay level which is SEK 500,000 (€55,000) according to the Swedish National Board of Health and Welfare.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Saghafi E, Kadhim K, Andas CA, Cahlin BJ, Finizia C, Axelsson T, Kjeller G, Tuomi L. Jaw exercise in head and neck cancer patients for prevention of temporomandibular disorders: a randomized controlled trial. J Cancer Surviv. 2024 Nov 22. doi: 10.1007/s11764-024-01717-w. Online ahead of print. PMID 39576571
- [Background] Petersson K, Finizia C, Pauli N, Tuomi L. Preventing radiation-induced dysphagia and trismus in head and neck cancer-A randomized controlled trial. Head Neck. 2025 Jan;47(1):159-174. doi: 10.1002/hed.27886. Epub 2024 Aug 1. PMID 39091121